CLINICAL TRIAL: NCT02858115
Title: Use of Mini-fluid Challenge for Fluid Responsiveness Prediction During One-lung Ventilation
Status: Completed | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-30
Record Dates: First submitted 2016-08-03; First posted 2016-08-08 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Acute Circulatory Failure During One-lung Ventilation Surgery

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- one lung ventilation lung: patients requiring one lung ventilation lung resection.
  Interventions: Other: Fluid challenge; Other: Trans-oesophageal echography

INTERVENTIONS:
Other: Fluid challenge — 100 ml of crystalloid was infused over 1-min
Other: Trans-oesophageal echography — an echocardiographic assessment at 1-min,

SUMMARY:
During thoracic surgery, an excessive use of fluid results in pulmonary complications. Dynamic fluid responsiveness predictors are not easily usable during one lung ventilation. The investigators hypothesized that the assessment by transesophageal echocardiography (TEE) of subaortic velocity time index (VTI) variation after 100 ml of crystalloid would predict fluid responsiveness in patients receiving one-lung ventilation.

This retrospective, observational, single center study was from January 2014 to December 2015. The investigators included 105 patients requiring one lung ventilation lung resection. The investigators analysed 39 patients presenting an acute circulatory failure. 100 ml of crystalloid was infused over 1-min. After an echocardiographic assessment at 1-min, remaining 400 ml were administered over 14-min Fluid responsiveness was defined as an increase in the VTI above 15% after infusion of 500 ml of crystalloid.

ELIGIBILITY:
Inclusion Criteria:

* Lung resection
* Acute circulatory failure
* One-lung ventilation

Exclusion Criteria:

* Sinusal rhythm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring one lung ventilation lung resection.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Fluid responsiveness | one day
  increase of cardiac output of more than 15%
Velocity time index | one day
  : Echographic assesment of cardiac output

SECONDARY OUTCOMES:
Pulsed pressure variation | one day
  dynamic indice of fluid responsiveness

CONTACTS AND LOCATIONS:
Locations (1):
- hôpital Nord Assistance Publique Hôpitaux de Marseille, Marseille, France